CLINICAL TRIAL: NCT07248319
Title: Production and Evaluation of an Evidence-based Health Awareness Video on Precautionary Measures Against Respiratory Infectious Diseases: A Randomized Controlled Trial on Public Transportation Drivers in Lebanon (HAV-RID Study)
Brief Title: Production and Evaluation of an Evidence-based Health Awareness Video on Precautionary Measures Against Respiratory Infectious Diseases (HAV-RID Study)
Acronym: (HAV-RID)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Mahmoud Salam, Assistant Professor, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LAU.SON.MS1.18/Dec/2025
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Produce and Evaluate an Evidence-based Health Awareness Video
Keywords: influenza; covid-19; transportation; health awareness video; Lebanon
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Intervention Model Description: After the video is produced, a non-blinded, randomized, two-arm controlled trial will be conducted. The experimental group will watch the newly produced health-awareness video, whereas the control group will watch a neutral video (raising awareness about traffic signs in Lebanon, https://www.youtube.com/watch?v=hb3107sylj0 ). The participants' knowledge about RID, health-risk perceptions, attitude towards vaccination, and cognitive dissonance will be evaluated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (n=80) will watch the health-awareness video (Experimental): The experimental group will watch the newly produced health-awareness video. Using a Delphi technique, the script will be revised by a panel of experts in public health, infection control, psychology, filmmaking, and public transportation (drivers, users, stakeholders). Experts will evaluate the script using two validated assessment tools, the Patient Education Materials Assessment Tool (PEMAT) and DISCERN. Once consensus is reached, the video will be produced.
  Interventions: Other: Health awareness video on precautionary measures against respiratory infectious disease
- control group will watch a neutral video (Active Comparator): control group will watch a neutral video (raising awareness about traffic signs in Lebanon, https://www.youtube.com/watch?v=hb3107sylj0 )
  Interventions: Other: Health awareness video on precautionary measures against respiratory infectious disease

INTERVENTIONS:
Other: Health awareness video on precautionary measures against respiratory infectious disease — Drafting of a narrative blueprint of the script for the health-awareness video is inspired by published and unpublished evidence-based studies previously conducted on public transportation drivers in Lebanon. This ensures the video content is evidence-based, culturally oriented, socially acceptable and tailored towards the target viewers. Using a Delphi technique, the script will be revised by a panel of experts in public health, infection control, psychology, filmmaking, and public transportation (drivers, users, stakeholders). Experts will evaluate the script using two validated assessment tools, the Patient Education Materials Assessment Tool (PEMAT) and DISCERN. Once consensus is reached, the video will be produced.

SUMMARY:
Health awareness videos are integral in disseminating knowledge about respiratory infectious diseases (RIDs). The aim of this study is to produce and evaluate an evidence-based health awareness video on precautionary measures against respiratory infectious diseases among public transportation drivers in Lebanon. You will be asked to watch a newly produced health-awareness video, then we will test your knowledge about respiratory infectious diseases , health-risk perceptions, attitude towards vaccination, and cognitive dissonance. Public transportation drivers are eligible to enroll if they operate within the Lebanese public transportation system, regardless of their gender. A proportionate sample of drivers will be invited to enroll from various Lebanese regions. The experimental group (n=80) will watch a health-awareness video, whereas the control group (n=80) will watch a neutral video on traffic signs. Participants' knowledge about RID, health-risk perceptions, attitude towards vaccination, and cognitive dissonance will be evaluated. The trial study will be conducted in community settings where public transportation drivers are naturally present (transportation stations, parking lots). A written informed consent will be sought. Data will be electronically recorded. Data will remain anonymous during data entry/analyses. An incentive will be provided.

DETAILED DESCRIPTION:
Background: Health awareness videos are integral in disseminating knowledge about respiratory infectious diseases (RIDs), elevating health-risk perceptions, and enhancing attitudes towards precautionary measures, as per the Health Belief Model (HBM) and Cognitive Dissonance Theory (CDT).

Aim: The aim of this study is to produce and evaluate an evidence-based health awareness video on precautionary measures against RID among public transportation drivers in Lebanon.

Methods: This project will be conducted over three stages and executed over two fiscal years (start date March 2026).

Stage one: Drafting the script of the video is inspired by seven published / unpublished evidence-based studies on public transportation drivers in Lebanon and fourteen studies from international literature. This ensures the video content is evidence-based, culturally oriented, socially acceptable and tailored towards the target viewers.

Stage two: Using a Delphi technique, the script will be revised by a panel of eight experts in public health, infection control, psychology, filmmaking, and public transportation using two validated assessment tools, the Patient Education Materials Assessment Tool (PEMAT) and DISCERN. A purposive sampling method will be followed. Once consensus is reached, the video will be produced.

Stage three: Non-blinded, randomized, two-arm controlled trial will be conducted by a group of senior nursing students (minimal risk study). Public transportation drivers are eligible to enroll if they operate within the Lebanese public transportation system, regardless of their gender. A proportionate sample of drivers will be invited to enroll from various Lebanese regions. Simple randomization technique will be performed. The experimental group (n=80) will watch the health-awareness video, whereas the control group (n=80) will watch a neutral video on traffic signs. Participants' knowledge about RID, health-risk perceptions, attitude towards vaccination, and cognitive dissonance will be evaluated. The trial study will be conducted in community settings where public transportation drivers are naturally present (transportation stations, parking lots). A written informed consent will be sought. Data will be electronically recorded. Data will remain anonymous during data entry/analyses. An incentive will be provided.

Data analysis: Data will be analyzed using SPSS; IBM (version 30). Knowledge statements will be scored and converted to percentage mean score. Risk perceptions, attitude and dissonance will be scored and converted to mean scores. Between group analyses of mean differences will be tested using student t-test and one way analysis of variance (ANOVA) with post hoc analysis (for normally distributed data) and Kruskall Wallis test with post hoc analysis (for skewed data). Forward stepwise linear regression analyses will be executed. Statistical significance will be at P<0.05 (two sided). Interim analysis will be performed at n=40.

Expected outcomes: Public transportation drivers and users might be unknowingly exposed to RID, so promoting their safety is a priority. When public transportation drivers are exposed to a video on RID, they will gain knowledge about it and demonstrate a positive attitude towards precautionary measures. This video contributes to higher service satisfaction and subsequently higher utilization of the transportation system. Utilizing the public transportation systems reduces street congestions, controls pollution, saves money for users and generates profits for stakeholders. Promoting a safe public transportation system reflects positively on public health, aligns with the CDC mission to control the global spread of diseases and lessens disease burden. Last but not least, health awareness videos are cost effective and they can reach a wider audience.

Ethical considerations: This study will not pose any risk or harm to participants. The video will not contain any material that might offend, insult, degrade, or discriminate against study participants in any way possible. Medical jargon and complex terms will be avoided. The video will be concluded with contact information in case participants decided to consult with experts in the future. Data collectors will be trained on how to remedy their concerns through cognitive behavioral therapy techniques to resolve negative thoughts, guide them on sources of knowledge and places to obtain facemasks, hand sanitizers and vaccines. Last but not least, participants will not be asked for any ID. The decision to participate or not will have no impact on drivers.

ELIGIBILITY:
Inclusion Criteria:

* Public transportation drivers who operate within the Lebanese public transportation system, regardless of their nationality or gender.

Exclusion Criteria:

* Commercial drivers (trucks) or others who are not in a daily contact with commuters.
* Drivers who are unwilling to enroll in the study or unable to comprehend written/verbal Arabic language will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 2 months
  Knowledge about RID mode of transmission and prevention will be evaluated (Khoury and Salameh 2015, Choucair, El Sawda et al. 2021). The percentage mean of knowledge scores (PMS±SD) will be presented. Higher scores indicate better knowledge. This variable measures the effectiveness of the health awareness video.
Patient Education Materials Assessment Tool - Audiovisual (PEMAT-AV) and • DISCERN tool | 5 months
  PEMAT-AV systematically evaluates the understandability and actionability of educational materials. Understandability is the viewers' ability to understand the video regardless of their diverse backgrounds and varying levels of health literacy. Actionability is the viewers' ability to identify what they can do based on the information presented in the video regardless of their background and level of health literacy. PEMAT produces separate numeric scores for understandability and actionability.
  DISCERN: to enable information providers to judge the quality of information about treatment choices. DISCERN facilitates the production of new, high quality, and evidence-based consumer health information. DISCERN became a reliable and valid instrument for judging the quality of written consumer health information.
Health-risk perceptions | 2 months
  Health-risk perceptions: participants' health-risk perceptions will be evaluated following two dimensions of the HBM that are the perceived susceptibility (2 items) and the perceived severity of RID (3 items) (Adams, Hall et al. 2014).
Attitude towards vaccination | 2 months
  participants' attitude towards vaccination will be evaluated using three domains of the Vaccination Attitudes Examination (VAX) scale: unexplored side effects of the vaccines (5 statements), pharmaceutical companies profiteering from vaccines (3 statements), and preferred reliance on natural immunity (3 statements). VAX is a generic tool that identifies people with negative attitudes towards vaccines (Martin and Petrie 2017).
Cognitive dissonance | 2 months
  dissonance is a self-reported measure of the emotional discomfort experienced due to cognitive dissonance (Elliot and Devine 1994). Cognitive dissonance can be measured using the dissonance thermometer that constitutes of adjectives distributed across four indices (discomfort index, negative self-index, shame index, and positive index). All four subscales demonstrated acceptable levels of reliability, with the positive and negative affect scales exhibiting excellent internal consistency and test-retest reliability (McGrath 2011). For this study, the discomfort index that constitutes of uncomfortable, uneasy, and bothered feelings will be used as adjective ratings (0 to 6). Higher score indicates an increased level of discomfort due to the effect of the video content.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Salam, PhD, Principal Investigator — Lebanese American University
Locations (1):
- Mahmoud Salam, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of IPD will follow local policies and regulations.

REFERENCES:
- [Result] Risk perceptions towards respiratory infectious diseases among university students utilizing the public transportation system in Lebanon
- [Result] Salam M, Haidar GH. Influenza vaccine hesitancy and its determinants among Lebanese public transportation drivers. Vaccine X. 2024 Dec 25;22:100606. doi: 10.1016/j.jvacx.2024.100606. eCollection 2025 Jan. PMID 39845631
- [Result] Exploring the Challenges that Public Transportation Drivers Face in Lebanon
- [Result] COVID-19 risk perceptions among public transportation drivers and users in Lebanon: A cross-sectional study